CLINICAL TRIAL: NCT04677036
Title: Self-Reported Surgeon Health Behaviours: A Multicentre, Observational Exploration With the Association of Surgeons in Training Into the Modifiable Factors That Impact Surgical Performance
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Dale Whelehan, Principal Investigator, University of Dublin, Trinity College
Record Dates: First submitted 2020-11-27; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TUH Staff: Staff within Tallaght University Hospital - anonymised
  Interventions: Other: No intervention is given
- ASIT Members: Members of the Association of Surgeons in Training - anonymised
  Interventions: Other: No intervention is given

INTERVENTIONS:
Other: No intervention is given — No intervention given
  Other Names: No intervention given

SUMMARY:
Introduction: Surgeons regularly educate patients on health promoting behaviours including diet, sleep and exercise. No study thus far has explored surgeons' personal compliance with these health-behaviours and their relationship with surgical performance.

The primary outcomes this study were self-reported health, health related behaviours, wellbeing, fatigue and surgical performance. Methods: A survey of validated themes on health-related behaviours, workplace variables and performance was distributed to surgical trainees and consultants in the UK and Ireland through the Association for Surgeons in Training (ASiT). Non-parametric analysis was used to determine inferential associations. Results: Ninety five surgeons (median age 35-44, 51.5 % female, 39.9% registrars) completed the survey. 94% reported having at least 'good' overall health. . A majority (54.7%) report inconsistent sleep patterns, while less than a quarter engage in regular exercise. 74% reported having at least 'good' overall mental and emotional well being.

Sixty two and 64.2% reported being regularly fatigued and bothered by feelings of anxiety and/or depression respectively. Poor self-reported health and wellbeing were associated with poorer reported off-call performance (p<.01). Higher levels of fatigue negatively impacted self-reported surgical and non-surgical task proficiency (p<.01). Discussion and Conclusion: Surgeons reported high levels of overall health. However, healthy behaviours around sleep, diet and exercise were not consistently reported. Fatigue, anxiety and regular rumination were reported by greater than half of respondents. When compared to overall health numbers, 20% less surgeons reported overall mental health and emotional well-being that good or better. Self-reported health behaviours including sleep and physical activity were associated with surgical performance. Strategies to improve modifiable lifestyle factors, which will optimise physical health, mental wellbeing and levels of fatigue may optimise surgical performance. Further research should target these behaviours to elicit desired changes.

ELIGIBILITY:
Inclusion Criteria:

* surgeon
* working in TUH or member of ASIT

Exclusion Criteria:

* non surgeon
* not a member of ASIT or TUH

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Trainees and consultant surgeons
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Self-reported health and wellbeing [This was a survey which was designed and validated as part of the study] | June-August 2020
  Likert scale:
  In general, how would you rate your overall health? In general, how would you rate your overall mental or emotional health? During the past 4 weeks, how disruptive were your physical health or emotional problems to your normal professional activities?
Levels of Fatigue | June-August 2020
  Likert Scale:
  In a typical week, how often do you feel fatigued at work?
  I manage work-related fatigue effectively.

SECONDARY OUTCOMES:
Sleep Outcomes | June-August 2020
  How many caffeinated drinks do you have each day? How often do you complete on-call work? How many hours do you sleep on average each night on a week without on-call? How many hours do you sleep on average each night on a week without on-call? How many hours on average do you sleep after on-call?
Performance Outcomes | June-August 2020
  In general, how would you rate your overall daily work performance when you're not on-call? In general, how would you rate your overall daily work performance when on-call? In a typical week, how often do you feel fatigue negatively impacts your ability to perform surgical tasks optimally?
Stress Outcomes | June-August 2020
  In a typical week, how often do you feel stressed at work? I find it easy to switch off after work.
Commuting Outcomes | June-August 2020
  How long do you typically spend commuting to work daily? How long do you typically spend commuting from work daily?
Physical Activity Outcomes | June-August 2020
  How many times in the average week do you engage in 30 minutes of light activity (i.e. leisurely walking, gardening, cleaning around the house)? How many times in the average week do you engage in 30 minutes of moderate activity (i.e. brisk walking, light bicycling)? How many times in the average week do you engage in 30 minutes of strenuous activity (i.e. running or jogging)? Do you feel you get too much exercise, too little exercise, or about the right amount of exercise?
Diet Outcomes | June-August 2020
  How often do you eat breakfast? How often do you eat lunch? How often do you eat dinner? How often do you eat fast food? How many portions of fruit do you eat each day? If you don't know for certain, please provide an estimate. How often do eat sweet things e.g. sweets, chocolate, crisps?
Health Check Outcome | June-August 2020
  When is the last time that you saw a doctor? When is the last time that you saw a dentist?
Work Culture Outcome | June-August 2020
  * In my experience, surgery staff are treated fairly when they make mistakes. We have enough staff to handle the workload.
  * Error disclosure is promoted and implemented effectively in our profession.
  * I have made major work-errors as a result of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Dale F Whelehan, BSc, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Tallaght University Hospital, Dublin, XX - Other State/Province/Territory, Ireland

IPD SHARING:
Plan to Share IPD: No